CLINICAL TRIAL: NCT05341505
Title: Outcomes and Neural Mechanisms of Emotion Regulation Therapy in Young Adults With Autism: A Pilot Feasibility Study
Brief Title: Outcomes of Emotion Regulation Therapy in Young Autistic Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michal Assaf (Other)
Responsible Party: Sponsor-Investigator, Michal Assaf, Director, Autism & Functional Mappin lab, Hartford Hospital
Organization: Hartford Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-HHC-2017-0161
Record Dates: First submitted 2022-03-24; First posted 2022-04-22 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Autism
Keywords: Emotion regulation
MeSH Terms: conditions — Autistic Disorder; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ER intervention (Experimental): Cognitive-behavioral emotion regulation intervention administered twice weekly for 8 weeks.
  Interventions: Behavioral: Emotion Regulation Intervention

INTERVENTIONS:
Behavioral: Emotion Regulation Intervention — We will administer a cognitive-behavioral treatment targeting emotion dysregulation, including mindfulness skills and other cognitive and behavioral emotion regulation skills.

SUMMARY:
This pilot study is designed to investigate the clinical outcomes and neural mechanisms of emotion regulation behavioral treatment , in a small sample of young adults diagnosed with autism spectrum disorder.

DETAILED DESCRIPTION:
Five young adults with ASD with emotional/behavioral challenges that are attributed to emotion dysregulation will be enrolled into an emotion regulation (ER) intervention administered twice weekly for a total of 16 sessions. Participants will be evaluated pre- and post-treatment using behavioral and imaging measures, and at mid-treatment and 2-month follow-up using behavioral measures administered electronically and/or via phone interview.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder
* Ages 18-40
* Estimated full-scale IQ ≥ 80
* T score > 60 on either the externalizing or internalizing symptoms scores of either the Adult Behavior Checklist (ABC-L) or the Adult Self Report (ASR)
* Participation in previous study at the Olin Center ("Social Emotional Study"; E-HHC- 2018-0241)

Exclusion Criteria:

* Intellectual disability (estimated full scale IQ<80
* History of a significant head injury (severe concussion, hospitalization)
* History of neurosurgery
* History of epilepsy, stroke, MS, a neurodegenerative disorder, or any other neurological disorder
* A current major medical condition (e.g. cancer, heart failure)
* Current substance use (determined by urine screen done to all participants before each MRI scan)
* In-body metal implants (e.g. surgical clips, certain pacemakers) or history of exposure to metal shards or other MRI contraindications
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Adult Self Report (ASR) | Baseline
  Externalizing and internalizing composite scores
Adult Self Report (ASR) | 8 weeks
  Externalizing and internalizing composite scores
Adult Self Report (ASR) | 2 months follow-up
  Externalizing and internalizing composite scores
Adult Behavior Checklist (ABC-L) | Baseline
  Externalizing and internalizing composite scores
Adult Behavior Checklist (ABC-L) | 8 weeks
  Externalizing and internalizing composite scores
Adult Behavior Checklist (ABC-L) | 2 months follow-up
  Externalizing and internalizing composite scores

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Living, Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No